CLINICAL TRIAL: NCT03666546
Title: Blood Glucose Response After Oral Intake of Lactulose (Laevolac®) in Mildly Constipated Patients With Diabetes Mellitus Type 2
Brief Title: Blood Glucose Response After Oral Intake of Lactulose in Mildly Constipated Patients With Diabetes Mellitus Type 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Lact-004-CP4; 2018-002359-14 (EudraCT Number)
Record Dates: First submitted 2018-08-23; First posted 2018-09-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Blood glucose; Diabetes Mellitus, Type 2; Lactulose; Constipation; Oral intake
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Constipation | interventions — Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Laevolac crystals 20 g (Experimental): Lactulose crystals, oral intake, 20 g single dose
  Interventions: Drug: Lactulose crystals 20 g
- Laevolac crystals 30 g (Experimental): Lactulose crystals, oral intake, 30 g single dose
  Interventions: Drug: Lactulose crystals 30 g
- Laevolac liquid 20 g (Experimental): Lactulose liquid, oral intake, 20 g single dose
  Interventions: Drug: Lactulose liquid 20 g
- Laevolac liquid 30 g (Experimental): Lactulose liquid, oral intake, 30 g single dose
  Interventions: Drug: Lactulose liquid 30 g
- Glucose 30 g (Active Comparator): Glucose Monohydrate, oral intake, 33 g single dose
  Interventions: Drug: Glucose
- Water (Placebo Comparator): Still water, oral intake, 250 mL single dose
  Interventions: Drug: Still water

INTERVENTIONS:
Drug: Lactulose crystals 20 g — White or almost white crystalline powder. The product will be provided in sachets to be dissolved in 250 mL water.
  Other Names: Laevolac crystals 20 g
  Arms: Laevolac crystals 20 g
Drug: Lactulose crystals 30 g — White or almost white crystalline powder. The products will be provided in sachets to be dissolved in 250 mL water.
  Other Names: Laevolac crystals 30 g
  Arms: Laevolac crystals 30 g
Drug: Lactulose liquid 20 g — Clear, viscous liquid, colourless or pale brownish-yellow liquid syrup (solution). The products will be provided in sachets to be dissolved in 250 mL water.
  Other Names: Laevolac liquid 20 g
  Arms: Laevolac liquid 20 g
Drug: Lactulose liquid 30 g — Clear, viscous liquid, colourless or pale brownish-yellow liquid syrup (solution). The products will be provided in sachets to be dissolved in 250 mL water.
  Other Names: Laevolac liquid 30 g
  Arms: Laevolac liquid 30 g
Drug: Glucose — White crystalline powder. To standardise for 30 g glucose, 33 g glucose monohydrate will be used. The products will be provided in sachets to be dissolved in 250 mL water.
  Other Names: Glucose Monohydrate
  Arms: Glucose 30 g
Drug: Still water — 250 mL still water will be used. Water from the same source will be also used to dissolve investigational and control products
  Other Names: Water
  Arms: Water

SUMMARY:
The objective of the study is to investigate whether lactulose, given orally as powder or liquid, increases blood glucose levels in patients with diabetes mellitus type 2. The dose of lactulose given in the study is normally used for treatment of constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-insulin requiring diabetes mellitus type 2 treated with diet and oral antidiabetics and/or Glucagon-like Peptide 1 receptor agonists
2. Age: 18-75 years
3. Female and male
4. Caucasian
5. HbA1c ≤ 7.5 %
6. Stable treatment, i.e. no change in diabetes mellitus related medication within the last 3 months
7. Mild functional constipation according to modified Rome IV criteria fulfilled for the last 3 months with symptom onset at least 6 months before study start defined as:

   * approx. 3-5 bowel movements per week,
   * of which 1-2 usually cause discomfort e.g., straining, lumpy or hard stools, sensation of incomplete evacuation or anorectal obstructions/blockage
8. Availability and presence in the trial unit for approx. 4 hours/ week for 4 weeks
9. Women of childbearing potential must be using a medically approved method of contraception OR women must be postmenopausal for at least 12 months prior to study entry
10. Signed informed consent form

Exclusion Criteria:

1. Fasting blood glucose <4.4 mmol/L (<80 mg/dL) or >10 mmol/L (>180 mg/dL) (capillary)
2. BMI <18.5 kg/m² or ≥35 kg/m²
3. Change in body weight ≥10 % within the last 3 months
4. Smoker
5. Major medical or surgical event requiring hospitalization within the last 3 months
6. Acute gastrointestinal diseases including diarrhea and/or vomiting within the last 2 weeks
7. Presence of disease or intake of drug(s) / supplements other than antidiabetic treatment influencing digestion and absorption of carbohydrates or bowel habits (intake of laxatives in general allowed with exception see next criterion) (dietary / supplementary fibres allowed if stable dose since 1 month before study start)
8. Not willing to abstain from laxatives 2 days before the visits 1-4 and up to 24h after visits 1-4
9. Use of following medication/ supplementation within the last 4 weeks and during the study:

   * Intake of medications other than antidiabetic treatment known to affect glucose tolerance e.g., steroids, protease inhibitors or antipsychotics;
   * Intake of prebiotics or probiotics
   * Chronic intake of substances affecting blood coagulation (e.g. acetylic acid (100 mg as standard prophylactic treatment allowed when dose is stable 1 month prior to screening), anticoagulants, diuretics, thiazides (diuretics and thiazides allowed e.g. for hypertension treatment when dose is stable 1 month prior to screening)), which in the investigator's opinion would impact patient safety
10. Severe liver, renal or cardiac disease
11. Hereditary problems of galactose or fructose intolerance, lactase deficiency or glucose-galactose malabsorption
12. Suspicion of alcohol abuse (defined as an average daily intake of more than one litre of beer per day or equivalent amount of alcohol in other beverages) or drug abuse
13. Known or suspected allergy to the investigational drug(s) or other components of the study drug(s)
14. Acute inflammatory bowel disease (ulcerative colitis, Crohn's disease), gastrointestinal obstruction or subocclusive syndrome, perforations or risk of perforation in gastrointestinal tract, abdominal pain of undetermined cause
15. Known history of human immunodeficiency virus (HIV), hepatitis B and/or C
16. Pregnancy, lactation
17. Clinically relevant findings as established by medical history, physical examination, clinical laboratory and/or vital signs
18. Participation in another interventional study with an investigational drug or an investigational medical device within 30 days prior to start of study or during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose levels as baseline corrected AUC: AUCbaseline_c (0-180 minutes) [Baseline corrected area under curve from 0 to 180 minutes for blood glucose concentration (= Area under curve from 0 to 180 minutes minus baseline*180 minutes)] | 0 - 180 minutes, during 4 study visits

SECONDARY OUTCOMES:
Maximum blood glucose concentration (Cmax) | 0 - 180 minutes, during 4 study visits
Maximum increase of blood glucose concentration (Max_increase) | 0 - 180 minutes, during 4 study visits
Relative maximum increase of blood glucose concentration (Max_increase_rel) | 0 - 180 minutes, during 4 study visits
Time to reach maximum blood glucose concentration (Tmax) | 0 - 180 minutes, during 4 study visits
Total area under curve from 0 to 180 minutes for blood glucose concentration (AUC(0-180 minutes)) | 0 - 180 minutes, during 4 study visits
Incremental area under curve from 0 to 180 minutes for blood glucose concentration, i.e., above baseline levels for blood glucose concentration after oral intake of Laevolac crystals/liquid or control products (iAUC(0-180min)) | 0 - 180 minutes, during 4 study visits

OTHER OUTCOMES:
Adverse Events (AEs) | up to 64 days
  Adverse Events will be documented from start of fasting on the day before Screening until the day after the last study Intervention. This is up to 64 days, depending on the day of Screening (21 to 3 days before the first study Intervention) and on the duration of wash out phases between interventions.
Gastrointestinal tolerability: global scaled evaluation | 180 minutes and 24 hours post-dose
  Gastrointestinal tolerability will be assessed by the patients by means of a global scaled evaluation with "Very good", "Good", "Moderate", or "Poor".
Gastrointestinal tolerability: diarrhoea, distension, rumbling, nausea, vomiting, burping, regurgitation/heartburn, flatulence, abdominal discomfort, abdominal pain | 180 minutes and 24 hours post-dose
  The single gastrointestinal symptoms will be assessed by the patients using a 4-point Likert scale: "No symptoms or discomfort", "Mild symptoms or discomfort", "Moderate symptoms of discomfort", or "Severe symptoms of discomfort".
Blood glucose concentration at 240 minutes - only when blood glucose is >10 mmol/L (>180 mg/dL) at 180 minutes | 240 minutes post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pieber, Prof. MD, Principal Investigator — Head and Chair of Department of Internal Medicine, Division of Endocrinology and Diabetology, Medical University, Graz, Austria
Locations (1):
- Clinical Research Center (CRC), Graz, Austria

IPD SHARING:
Plan to Share IPD: No